CLINICAL TRIAL: NCT07237737
Title: Wound Healing Outcomes With and Without the Alexis Wound Retractor in Direct Anterior Approach Total Hip Arthroplasty
Brief Title: Alexis Retractor in Total Hip Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Professor of Orthopaedic Surgery, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20251013
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hip Osteoarthritis; Hip Arthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Alexis Retractor (Experimental): Subjects in this arm will undergo surgery using the Alexis wound retractor.
  Interventions: Device: Alexis wound retractor
- Non-Alexis Retractor (Active Comparator): Subjects in this arm will undergo surgery using a standard retractor that does not include the Alexis device.
  Interventions: Device: Standard wound retractor

INTERVENTIONS:
Device: Alexis wound retractor — A surgical device used to retract tissue during procedures, designed to reduce wound trauma and improve healing
  Arms: Alexis Retractor
Device: Standard wound retractor — A conventional surgical retractor used during procedures without the features of the Alexis device
  Arms: Non-Alexis Retractor

SUMMARY:
To determine if there is a difference in wound healing and surgical site infection (SSI) rates using the Alexis wound retractor vs. not using it in longitudinal direct anterior approach total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral longitudinal direct anterior approach total hip arthroplasty
* Patients undergoing primary total hip arthroplasty

Exclusion Criteria:

* Patients with history of prior open surgery on the affected hip
* Patients with history of prior total hip arthroplasty on the contralateral hip
* Patients with allergies or absolute contraindication to standardized drugs administered within the University of Miami protocol for total hip replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of Days to Identification of Delayed Wound Healing | Up to 14 days
  Delayed wound healing is defined as the presence of one or more of the following clinical signs: drainage from wound, wound dehiscence, and superficial surgical site infection. Assessment is performed by clinical examination and documentation in the postoperative period. The outcome is measured in number of days from surgery to identification of delayed healing
Patient satisfaction with scaring as measured by Patient Scar Assessment Scale | Up to 12 months
  Using the Patient Scar Assessment Scale, which is a validated plastic surgery tool for evaluating scars from the patient's perspective. Measured with a scale from 0 to 10, higher score indicates less satisfaction.
Scar cosmesis as measured by Observer Scar Assessment Scale | Up to 12 months
  Using the Observer Scar Assessment Scale, which is a validated plastic surgery tool for evaluating scars from the observer perspective. Measured with a scale from 0 to 10, higher score indicates worse scar cosmesis.

SECONDARY OUTCOMES:
Number of Participants Reporting Lateral Femoral Cutaneous Nerve (LFCN) Symptoms | Up to 6 months
  LFCN symptoms are defined as paresthesias or dysesthesias in the anterior thigh distal to the surgical site. Symptoms are assessed through participant self-report and clinical documentation.
Hip Disability and Osteoarthritis Outcome Score (HOOS) - Patient-Reported Outcome | Up to 12 months
  Assessed using the HOOS, a validated instrument for evaluating hip-related disability and osteoarthritis symptoms from the patient's perspective. Scores range from 0 to 28, with higher scores indicating worse patient-reported outcomes.
Number of Intraoperative fractures | Up to 3 hours (duration of surgery)
  Intraoperative complications will be assessed by counting the number of fractures occurring during the surgical procedure; fractures are identified by the operating surgeon and confirmed via intraoperative imaging or direct visualization.
Length of surgery | Up to 3 hours
  Duration of the surgical procedure measured in minutes, from initial incision to closure.
Number of Postoperative Complications | Up to 90 days
  Measured by the number of complications including, but not limited to, periprosthetic joint infection (PJI), prosthetic hip dislocation, periprosthetic fracture, implant failure requiring revision surgery. Events are identified through clinical evaluation and documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Victor H Hernandez, MD, MSc, Principal Investigator — University of Miami Department of Orthopaedics
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No